CLINICAL TRIAL: NCT06473714
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Inhibition and Brain Function in Primary Progressive Aphasia
Acronym: Stim-APHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-AOI-07
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Aphasia, Primary Progressive
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS (Experimental)
  Interventions: Device: tDCS
- SHAM (Sham Comparator)
  Interventions: Device: SHAM

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation of the dorsolateral prefrontal cortex will be made at 1,5mA
  Arms: tDCS
Device: SHAM — Transcranial direct current stimulation of the dorsolateral prefrontal cortex will not be made. The electrodes are placed on the skull and a slight but non-continuous intensity is applied.
  Arms: SHAM

SUMMARY:
Primary progressive aphasia (PPA) is a focal dementia characterized by primary impairment of language abilities and functional disturbances associated with language.

Although PPA is a progressive disorder, new techniques are being proposed to try to activate parts of the brain previously thought to be potentially inactive, due to the possibility of "neuroplasticity". This concept refers to our brain's modularity and learning potential. Transcranial direct current stimulation is a powerful neuromodulatory technique, in which a small current is applied to the participant's scalp through the targeted positioning of an anode and a cathode. The positive or anodal stimulation of tDCS is supposed to increase neuronal activity under the electrode, while cathodal stimulation is supposed to do the opposite.

This project will provide new insights into the nature of the neural activity underlying executive functions in people with primary progressive aphasia compared to those without. The investigators expect to find reduced amplitude of electrophysiological responses and lower accuracy in people with primary progressive aphasia compared with healthy controls. Given the results of previous studies showing the efficacy of tDCS protocols in the treatment of aphasia, the investigators might expect them to improve executive functions. If so, the investigators expect significantly greater electrophysiological responses after stimulation sessions compared with sham conditions. This project is of great clinical relevance. This research will improve current therapeutic protocols used in the treatment of PPA by providing critical findings on whether and how the use of tDCS improves executive functions. Crucially, the research will advance knowledge of executive function decline as a sensitive marker of PPA, informing us about the possibility of early detection of this disorder. At the same time, the investigators will analyze the possibility of controlling symptomatological evolution via the analysis of acoustic and vocal markers. This will enable us to observe the evolution of sensory markers such as acoustic markers according to symptomatological evolution. This will enable us to check whether acoustic markers correlate with the patient's level of symptomatological impairment and/or pathological physiological data.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female over the age of 18 with a primary progressive aphasia diagnosis
* Available for treatment and testing sessions
* able to read and speak French
* Be right-handed

Exclusion Criteria:

* Presence of neurodevelopmental disorders or non-degenerative neurological disorders
* Post-stroke aphasia
* Language or cognitive disorders too severe to allow task performance or communication
* Pre-existing psychiatric disorders; severe depression, schizophrenia
* People with pacemakers or metal implants, epilepsy
* Presence of a medical condition that represents a contraindication to tDCS
* Active use of psychotropic drugs
* Treatment with tDCS or TMS in the last 3 months
* Additional language therapy
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Flanker task | 6 week
Stroop task | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Auriane Gros, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No